CLINICAL TRIAL: NCT00808522
Title: Prevention of Breast Cancer: As Simple as hCG-A Randomized Clinical Trial in High Risk Women.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Giuseppe Del Priore, New Downtown Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GD-10-08
Record Dates: First submitted 2008-12-13; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Chemoprevention; Tamoxifen; Breast density; Hcg
MeSH Terms: conditions — Breast Neoplasms; Hypertrichosis congenital generalized X-linked

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hCG (Experimental): Patients at high risk for breast cancer will be treated with hCG
  Interventions: Drug: hCG
- routine care (No Intervention): Patients receiving routine care will be followed
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: hCG — recombinant hCG subcutaneous injections x 30 doses every other day lasting 60 days total.
  Other Names: Ovidril

SUMMARY:
The purpose of the study is to evaluate whether hCG will result in a decrease in breast density.

High breast density has been associated with an increased risk in breast cancer. It has also been shown that decreasing density with a drug called tamoxifen has resulted in a decreased risk in breast cancer. The investigators are looking at the effect of hCG on breast density in people who are at increased risk of developing breast cancer and our theory postulates that through the hormonal actions of hCG and tamoxifen there would be a greater reduction in breast density in patients who are treated with hCG and tamoxifen versus patients treated with tamoxifen alone. Using this data the investigators will be able to hypothesize that the treatment of hCG will result in a reduction in breast cancer rates in the population and thus make available another drug which can be used to decrease the rates of breast cancer in the population

DETAILED DESCRIPTION:
Pregnancy has been associated with a decreased risk of breast cancer. This has been reproduced in multiple studies and has been seen in multiple races.

People have been evaluating different hormones and practices associated with pregnancy to determine what factors reduce the risk of developing breast cancer in these patients. These pronounced findings have been evaluated in great detail by multiple scientists and one of the hormones which we think might be associated with a reduction in breast cancer is hCG. This statement has been backed by multiple studies which have looked at the direct effect of hCG on the growth and death of breast cancer cells in the lab and in animal models of breast cancer.

We want to determine if hCG is given to patients who are at increased risk of breast cancer will result in an accentuated decrease in breast cancer risk above and beyond the effect received by conventional breast cancer reducing protocols. Our final outcome in this study will be breast density on mammographic evaluation which is considered a marker for breast cancer. So our study will evaluate whether or not hCG will have an effect on the mammographic breast density.

After recruitment there will be two groups in our study an intervention group and non intervention group. In the intervention group patients would undergo a period of hCG injections which would last a total of 60 days and consist of 30 subcutaneous injections. The non intervention group will continue their conventional chemoprevention medication. Both groups will be followed for teo years and the images, cytology and blood samples will be sent to our labs for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* On tamoxifen therapy for the treatment or prevention of breast cancer.
* Must have at least one remaining breast.

Exclusion Criteria:

* Pregnant or nursing.
* No history of allergic reactions to hCG.
* Patients who have had bilateral mastectomies.
* Uncontrolled thyroid disease.
* Cognitively impaired and unable to consent for the trial.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The investigators will be looking at the mammographic breast density at the start of the trial and then every 6 months for 2 years. The treatment arm will have 30 injections of Hcg over a 60 day period. | 2 years

SECONDARY OUTCOMES:
Evaluation of breast cytology and serum hormone levels at 6 monthly intervals over the course of the study. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- New York Downtown Hospital, New York, New York, United States